CLINICAL TRIAL: NCT05725135
Title: Gender Differences in Propofol Requirements During Total Intravenous Anaesthesia Administered by Closed-loop Anaesthesia Delivery System: An Observational Study
Brief Title: Effect of Gender on Propofol Requirement
Status: Completed | Type: Observational
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Nitin Sethi, DNB, Senior Consultant, Sir Ganga Ram Hospital
Other Study IDs: EC/01/23/2217
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Anesthesia
Keywords: propofol; male; female
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Males: Propofol total intravenous anaesthesia (TIVA) will be used for both induction and maintenance of anaesthesia. Propofol administration rate will be controlled by a feedback loop facilitated by BIS monitoring using automated closed-loop anesthesia delivery system (CLADS). A BIS value of 50 will be used as the target point for induction and maintenance of anaesthesia.
  Interventions: Drug: Propofol
- Females: Propofol total intravenous anaesthesia (TIVA) will be used for both induction and maintenance of anaesthesia. Propofol administration rate will be controlled by a feedback loop facilitated by BIS monitoring using automated closed-loop anesthesia delivery system (CLADS). A BIS value of 50 will be used as the target point for induction and maintenance of anaesthesi
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Propofol total intravenous anesthesia (TIVA) will be used for induction and maintenance of anesthesia. Propofol will be delivered using automated closed-loop anesthesia delivery system.

SUMMARY:
Total intravenous anaesthesia (TIVA) has emerged as a viable alternative to inhalational general anaesthesia (GA). Propofol is the preferred drug for providing TIVA due to its favorable pharmacokinetic profile, such as, rapid onset of action and a short context sensitivity half -life. There is suggestion that consumption of Propofol required during TIVA is influenced by gender with females requiring higher dose due to higher volume of distribution of drug. The evidence on gender differences in Propofol requirement for TIVA is largely based on studies done using subjective (manual titration of infusions)/semi-objective (target-controlled infusions) methods of drug administration, whose initial setting and ongoing control may be affected by attending anesthesiologist discretion and action. A recent advance in Propofol TIVA delivery is development of objective automated anaesthesia delivery systems. These systems administer Propofol titrated to patients' electroencephalogram (EEG) response reflected by processed EEG monitoring, namely the Bispectral index (BIS). One such indigenously developed automated anaesthesia delivery system is the closed-loop anaesthesia delivery system (CLADS). CLADS is a more precise and robust system to facilitate administration of Propofol TIVA, which automatically regulates the dose of medication based on feedback from patient's BIS data. The present study proposes to explore if there can be any gender differences in Propofol requirements during total intravenous anaesthesia administered by CLADS. All patients undergoing elective surgery under Propofol TIVA using CLADS will be screened, and those eligible will be enrolled. Enrolled patients will receive automated Propofol TIVA using CLADS. Demographic and clinical details including gender of patient will be noted. Cumulative dose of Propofol use will be computed through algorithm executed and monitored by software built into the CLADS. The findings will then be compared between male and female gender. Other intraoperative and post- operative outcomes such as time-to-loss of consciousness, time-to-induction of anaesthesia, anaesthesia depth consistency, performance characteristic of CLADS, hemodynamic profile (heart rate, mean arterial blood pressure), time-to-early recovery from anaesthesia, and postoperative sedation scale (modified observers' assessment of alertness/sedation scale [MOAA/S]); will be noted and compared between males and females. We expect to enroll 80 patients in our study.

DETAILED DESCRIPTION:
Total intravenous anaesthesia (TIVA) has emerged as a viable alternative to inhalational general anaesthesia (GA). Progress into TIVA is much desirable for continued development of precision GA. To this effect, Propofol is a key intravenous agent because of its favorable pharmacokinetic (PK) and pharmacodynamic (PD) profile and broad administration applicability with different methods of delivery: manual and target-controlled infusion [TCI].

The evidence on gender differences during manual/TCI Propofol TIVA suggests that females as compared to males have increased requirement of Propofol and yet have a faster time to recovery from anaesthesia. A 5-10% excess body fat and 15-20% decreased water content in females as compared to males' results in an increase in volume of distribution (Vd) of lipophilic drugs (e.g., Propofol), which consequently necessitates a higher rate of delivery of the Propofol infusion to achieve the same plasma concentration (as males) for clinically acceptable depth-of-anaesthesia. Whereas an increased Propofol sensitivity results in early awakening from anaesthesia.

The studies on gender differences in Propofol requirements and recovery from anaesthesia are largely based on semi-objective methods of Propofol TIVA administration (manual/TCI). The human element in titration and control of manual/TCI delivery of Propofol TIVA in above studies may be a limiting and a confounding factor in interpretating the actual difference induced by the 'gender' context. Whilst processed electroencephalogram (EEG) monitoring (Bispectral index [BIS], entropy, Narcotrend®) facilitates control of Propofol TIVA; it may still be imprecise due to subjective differences in understanding and execution of Propofol TIVA.

A recent advance in Propofol TIVA delivery is the development of automated anaesthesia delivery systems such as closed loop anaesthesia delivery system (CLADS). These systems administer Propofol actuated, titrated, and controlled by patients' processed electroencephalogram (EEG) response as generated by continuously monitored bispectral index (BIS) score. Current evidence suggests that automated Propofol TIVA delivery systems such as closed loop anaesthesia delivery system (CLADS) facilitate precision administration of Propofol than its TCI/manual counterparts.

Despite a plethora of evidence on effectiveness of Propofol TIVA, gender differences in Propofol PK and PD have not been evaluated while using automated systems of delivery. With the premise that widely researched and precise automated closed-loop anaesthesia delivery system (CLADS) has clear advantages (lower 'operator' dependence and inclusion of 'patient' factor) over manual/TCI mode; it is likely that Propofol TIVA administered by CLADS will lend greater objectivity in qualifying and quantifying the inter-gender differences in Propofol consumption and recovery from anaesthesia. The proposed observational study is planned to explore the gender differences in Propofol consumption and recovery from anaesthesia following CLADS controlled Propofol TIVA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years.
* ASA physical status I and II.
* Patients undergoing elective surgeries of minimum 1 hour duration.

Exclusion Criteria:

* Uncompensated cardiovascular disease (e.g., uncontrolled hypertension, systolic and diastolic dysfunction)
* Hepatic dysfunction (liver enzymes > 2 times the normal range)
* Renal dysfunction (serum creatinine > 1.4 mg/dl)
* Psychiatric or neurological disorder
* Uncontrolled endocrinology disease (diabetes mellitus, hypothyroidism)
* Known allergy/hypersensitivity to the study drug
* History of recent intake of sedative medication or anti-psychotic medication
* Drug dependence/substance abuse
* Requirement of postoperative ventilation
* Refusal to informed consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients undergoing elective surgery requiring general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Cumulative Propofol consumption (mg/kg/h) during anaesthesia | From start of Propofol injection 10-hours intraoperatively]
  Dose of Propofol required for induction and maintenance of anesthesia

SECONDARY OUTCOMES:
Time to loss of consciousness | From start of anesthesia till 5- minutes intraoperatively
  The time taken from starting Propofol induction using closed-loop anaesthesia delivery system till loss of verbal response will be recorded
Time to induction of anaesthesia | From start of anesthesia till 5- minutes intraoperatively
  The time taken from starting Propofol induction using closed-loop anaesthesia delivery system till a target BIS value of '50' is achieved
Intra-operative heart rate (beats per minute) | From beginning of anesthesia till 10 hours intraoperatively
  Comparison of intra-operative heart rate between the cohort groups will be done
Intra-operative systolic , diastolic, and mean blood pressure (mmHg) | From beginning of anesthesia till 10 hours intraoperatively
  Comparison of intra-operative blood pressure- systolic, diastolic, and mean blood pressure between the cohort groups will be done
Anesthesia depth consistency | From beginning of anesthesia till 10 hours intraoperatively
  It will be determined by the percentage of the anaesthesia time during which the BIS remained +/- 10 of the target BIS of 50
Performance characteristic of Propofol delivery system | From beginning of anesthesia till 10 hours intraoperatively
  It will be determined using the Varvel criteria parameter :median performance error (MDPE). This parameter is calculated by the computer software which analyses the intraoperative BIS data. This parameter have no unit of measurement. Its just a abstract number
Performance characteristic of Propofol delivery system | From beginning of anaesthesia till 10 hours intraoperatively
  It will be determined using the Varvel criteria parameter: median absolute performance error (MDAPE).This parameter is calculated by the computer software which analyses the intraoperative BIS data. This parameter have no unit of measurement. Its just a abstract number.
Performance characteristic of Propofol delivery system | From beginning of anaesthesia till 10 hours intraoperatively
  It will be determined using the Varvel criteria parameter: wobble. This parameter is calculated by the computer software which analyses the intraoperative BIS data. This parameter have no unit of measurement. Its just a abstract number.
Performance characteristic of Propofol delivery system | From beginning of anaesthesia till 10 hours intraoperatively
  It will be determined using the Varvel criteria parameter: global score. It is calculated using the formula Median absolute performance error + wobble / percentage of the anesthesia time during which the BIS remained +/- 10 of the target BIS of 50. This parameter have no unit of measurement. Its just a abstract number.
Early recovery from anesthesia | From end of anaesthesia till 20-minutes postoperatively
  Time taken by the patient to open his/her eyes after discontinuation of anaesthesia will be noted
Early recovery from anesthesia | From end of anaesthesia till 20-minutes postoperatively
  Time taken for tracheal extubation after discontinuation of anaesthesia will be noted
Postoperative sedation | From end of anaesthesia till 24-hours postoperatively
  Will be assessed using Modified Observer's assessment of alertness/sedation scale. The scale has a maximum value of '5', which refers to a fully awake patient and a minimum value of '0' which refers to a deeply sedated patient.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Sethi, DNB, Principal Investigator — Sir Ganga Ram Hospital, New Delhi, INDIA; Amitabh Dutta, MD, PGDHR, Study Director — Sir Ganga Ram Hospital, New Delhi, INDIA; Jayashree Sood, MD, FFRCA, PGDHHM, FICA, Study Chair — Sir Ganga Ram Hospital, New Delhi, INDIA
Locations (1):
- Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi, India